CLINICAL TRIAL: NCT03711981
Title: Laparoscopically Assisted Transversus Abdominis Plane Block Using Liposomal Bupivacaine and Laparoscopic or Robotic Gynecology: A Randomized Controlled Trial (#2)
Brief Title: Laparascopic TAP and Hysterectomy Trial #2
Acronym: TAP2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tennessee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16-027
Record Dates: First submitted 2018-05-02; First posted 2018-10-19 (Actual); Last update posted 2018-10-19 (Actual); Status verified 2018-05

CONDITIONS: Anesthesia
Keywords: laparascopic, surgery, anesthesia

STUDY DESIGN:
Intervention Model Description: Patients in one arm of the study would receive a bilateral Laparoscopic Assisted TAP block with 10cc Liposomal bupivacaine, 10cc 0.25% bupivacaine and 10cc normal saline each bilaterally at the beginning of their surgery. The patients in the control arm of the study would receive pre-incisional injections at the trocar incision sites using a total of 20cc 0.25% bupivacaine.
Who Masked: Participant
Masking Description: Participants will not know which type of injection they have received for pain control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAP block of 10cc Liposomal bupivacaine (Active Comparator): Patients in this arm of the study would receive a bilateral Laparoscopic Assisted TAP block with 10cc Liposomal bupivacaine, 10cc 0.25% bupivacaine and 10cc normal saline each bilaterally at the beginning of their surgery.
  Interventions: Procedure: TAP Block
- Routine pre-incisional injections at trocar incision sites (No Intervention): The patients in the control arm of the study would receive routine pre-incisional injections at the trocar incision sites using a total of 20cc 0.25% bupivacaine.

INTERVENTIONS:
Procedure: TAP Block
  Arms: TAP block of 10cc Liposomal bupivacaine

SUMMARY:
More than 600,000 hysterectomies are performed in the United States each year, making it the most common non-obstetric major surgery performed on women1. Estimates suggest that at least 30% of hysterectomies are performed laparoscopically or robotically with an increasing trend toward minimally invasive approaches2. While a minimally invasive approach certainly provides improved recovery, patients still experience substantial pain and most require opiate medications for pain control. Incorporating a multimodal approach to postoperative pain management through the use of field nerve blocks is potentially an ideal way to enhance recovery and minimize the need for narcotic pain medications.

Over the past decade, the use of Transversus Abdominis Plane (TAP) blocks as an adjunct for postoperative pain management has gained in popularity. First described in 2001 by Dr. Rafi of Limerick3, Ireland, TAP blocks are now typically performed by an anesthesiologist with the use of ultrasound guidance. The transversus abdominis plane is the neurovascular plane between the aponeurosis of the internal oblique and transversus abdominis muscles. Herein lie the afferent nociceptor nerve endings of T7-L1. Injection of a 20-30cc volume of anesthetic into this plane causes a sensory nerve block to the ipsilateral antero-abdominal wall from the costal margin to the symphysis pubis4.

Clinical trials have documented the validity of using TAP blocks for both open and laparoscopic procedures and verified their use for postsurgical pain relief. Studies have demonstrated that TAP blocks for both open and laparoscopic hysterectomies are safe and efficacious5, 6. In 2011, De Oliveira et al. demonstrated improved quality of recovery for women undergoing preoperative ultrasound guided TAP infiltration with ropivacaine at the time of laparoscopic hysterectomy7.

DETAILED DESCRIPTION:
The primary goal of our study is to demonstrate that laparoscopically assisted bilateral Transversus Abdominis Plane (TAP) block using liposomal bupivacaine is superior to pre-incisional injection of bupivacaine in terms of peri-operative opiate use, pain scores and overall patient satisfaction up to one week following surgery. Our recent research has already demonstrated the safety of performing Laparoscopic assisted TAP blocks using liposomal bupivacaine.

This trial will evaluate the efficacy of laparoscopic TAP blocks with liposomal bupivacaine by using VAS/numeric pain scores at rest and with cough in recovery at 1 and 2 hours post-op. The trial will also utilize an OBAS patient survey, document peri-operative opioid pain medication used intraoperatively, in PACU and overnight (if admitted), and assess length of time in PACU and same-day discharge versus admission. Opioid pain medication use at home up to one week will also be recorded.

HYPOTHESES/SPECIFIC AIMS The goal of this research project is to prove that a laparoscopically delivered TAP block using a combination of Liposomal bupivacaine (Exparel) and Bupivacaine is an effective and feasible means for decreasing post-operative pain from the immediate post-operative period up to one week.

The research aims to demonstrate that TAP blocks, when delivered laparoscopically and by using Liposomal bupivacaine will show a 20% benefit in post-operative QoR-15 scores on post-operative days 1,2 and 7. Other objectives of our study will be to evaluate peri-operative narcotic medication dosing, VAS/Numeric pain scores with cough at 1 and 2 hours in PACU, overnight narcotic use for patients who are admitted and narcotic pain pill use at home up to 7 days. Finally, the study aims to confirm that this technique is simple to perform, easy to implement and would offer a multi-modal anesthetic alternative to the excessive use of post-operative opioid pain medications.

Patients scheduled for laparoscopic or robotic hysterectomy are screened in the pre-anesthesia care unit and if eligible are invited to enroll in the trial. Primary Attendings for each surgery will advise patients of the option for the trial at pre-operative appointments. Patients who agree to enrollment are appropriately consented and then randomized to either control (pre-incisional anesthetic) or study (TAP) group. The patient remains blinded to the arm of the study, but OR personnel are advised so as to prepare medications and syringes.

Following induction of anesthesia, the patients in the TAP block arm are prepared and draped for surgery allowing for mid-axillary access along the flank bilaterally. Once pneumoperitoneum and a port for the laparoscope were established, TAP block is performed bilaterally by first palpating the external landmark within the Triangle of Petit, 2 cm above the iliac crest. A 21-gauge Stimuplex ® A insulated needle (Braun, Melsungen, Germany) is used to enter the transversus abdominis neurovascular plane. Bilaterally, TAP block patients receive 10cc of liposomal bupivacaine combined with 10cc of 0.25% bupivacaine and 10cc normal saline. Patients in the pre-incisional injection arm of the study receive a total of 20cc of 0.25% bupivacaine total, equally distributed between the incisions. All patients receive routine general anesthesia with opiate use adjusted as determined by the anesthesia provider. The anesthesia team is neither blinded nor given specialized protocol instructions. At the end of each case, narcotic dosage used is documented.

All of the patients will receive phone calls on post-operative days 1,2 and 7. They will be asked their opiate pain medication usage, number of pills used and "Overall Benefit of Anesthesia" (OBAS) scores will be obtained. The OBAS is a simple quality assessment instrument shown to reliably measure benefit from post-operative pain therapy16 (Table 1).

Table 1. Overall Benefit of Analgesia Score

1. Please rate your current pain at rest on a scale between 0=minimal pain and 10=maximum imaginable pain
2. Please grade any distress and bother from vomiting in the past 24 h (0=not at all to 10=very much)
3. Please grade any distress and bother from itching in the past 24 h (0=not at all to 10=very much)
4. Please grade any distress and bother from sweating in the past 24 h (0=not at all to 10=very much)
5. Please grade any distress and bother from freezing in the past 24 h (0=not at all to 10=very much)
6. Please grade any distress and bother from dizziness in the past 24 h (0=not at all to 10=very much)
7. How satisfied are you with your pain treatment during the past 24 h (0=not at all to 10= very much)

   OBJECTIVES The primary goal of our study is to demonstrate that laparoscopically assisted bilateral Transversus Abdominis Plane (TAP) block using liposomal bupivacaine is superior to pre-incisional injection of bupivacaine in terms of peri-operative opiate use, pain scores and overall patient satisfaction up to one week following surgery. Our recent research has already demonstrated the safety of performing Laparoscopic assisted TAP blocks using liposomal bupivacaine.

   This trial will evaluate the efficacy of laparoscopic TAP blocks with liposomal bupivacaine by using VAS/numeric pain scores at rest and with cough in recovery at 1 and 2 hours post-op. The trial will also utilize an OBAS patient survey, document peri-operative opioid pain medication used intraoperatively, in PACU and overnight (if admitted), and assess length of time in PACU and same-day discharge versus admission. Opioid pain medication use at home up to one week will also be recorded.

   HYPOTHESES/SPECIFIC AIMS The goal of this research project is to prove that a laparoscopically delivered TAP block using a combination of Liposomal bupivacaine (Exparel) and Bupivacaine is an effective and feasible means for decreasing post-operative pain from the immediate post-operative period up to one week.

   The research aims to demonstrate that TAP blocks, when delivered laparoscopically and by using Liposomal bupivacaine will show a 20% benefit in post-operative QoR-15 scores on post-operative days 1,2 and 7. Other objectives of our study will be to evaluate peri-operative narcotic medication dosing, VAS/Numeric pain scores with cough at 1 and 2 hours in PACU, overnight narcotic use for patients who are admitted and narcotic pain pill use at home up to 7 days. Finally, the study aims to confirm that this technique is simple to perform, easy to implement and would offer a multi-modal anesthetic alternative to the excessive use of post-operative opioid pain medications.

   PRELIMINARY WORK IRB protocol #14-132 was discontinued 12/14/15 due to a protocol violation. Because the study could not be completed with its original objectives, we are seeking to repeat the study with a very similar protocol. While talking with patients during the audit of their post-operative phone calls, it became clear that the experimental arm of the study might, in fact, have had a beneficial impact on post-operative recovery. As we do not have that portion of the data, we are seeking to repeat the study with a few minor modifications.

   METHODS
   1. Study Design Proposed study design is for a Prospective Single blinded Randomized Clinical Trial. The study aims to evaluate two arms and compare them: All patients would undergo laparoscopic total hysterectomy or Robotic assisted laparoscopic total hysterectomy with or without removal of adnexa. Patients would not be excluded for having other simultaneous procedures such as appendectomy, excision of endometriosis or pelvic lymph node dissection. Patients in one arm of the study would receive a bilateral Laparoscopic Assisted TAP block with 10cc Liposomal bupivacaine, 10cc 0.25% bupivacaine and 10cc normal saline each bilaterally at the beginning of their surgery. The patients in the control arm of the study would receive pre-incisional injections at the trocar incision sites using a total of 20cc 0.25% bupivacaine.
   2. Study Subjects

   <!-- -->

   1. Women undergoing laparoscopic hysterectomy or robotic assisted laparoscopic hysterectomy with or without removal of adnexa would be eligible. Patients will be randomized.
   2. Inclusion Criteria: Women undergoing TLH at Erlanger Hospital. They must be 18 years or older due to restrictions on Exparel. Women undergoing simultaneous lymph node dissection, appendectomy, adhesiolysis or other incidental procedures would not be excluded.
   3. Exclusion Criteria: Patient refusal. Soft tissue infection of the abdominal wall and skin. Abnormality at the needle insertion site. Chronic opiate use within 3 months prior to surgery. Age less than 18 years. Anticipated need for extension of incision greater than 2cm. Hepatic or renal impairment, current pregnancy or BMI >50.

   c. Sample Size: 100 patients, 50 in each arm of the study. The sample size calculation is based on an assumption that a 24% difference in VAS pain scores would be clinically meaningful. A sample size of 41 patients in each cohort would be able to detect a 20% difference in post-operative QoR-15 quality of life post-surgery scores with a power of 80%. This calculation was done with the assistance of Jenny Holcomb, PhD (See accompanying paperwork).

   d. Data Collection: Each patient will have paperwork designating name, demographics, telephone numbers as well as pertinent PHI. Documentation of VAS scores, time-frame to first request for opiate pain medications, post-operative pill counts and follow-up phone questionnaire (OBAS) will be collected on accompanying forms.

   e. Data Handling: A file, with the paper work on each patient, will be handled by the Principal Investigator, Shanti Mohling, MD and primary Co-investigator, Rayan Elkattah, MD. Two personnel will be recruited to handle post-operative phone calls. They will be carefully screened for reliability and phone-calls assessments will be periodically audited to avoid the concerns occurring with #14-132. The charts will be stored in the primary investigator's private office or in the research specialist's office (Patricia Bush) during analysis.

   f. Data Analysis: Following collection of data and collation of all data, the results will be statistically analyzed with the help of statistician Jenny Holcomb, PhD.

   g. Time Frame:

1. 12 months for data collection. 2. 18 months time for completion of study including analysis. h. Strengths/Innovation: Adding a simple technique for post-operative pain control to the armamentarium of multi-modal anesthesia techniques will greatly enhance the options for caring for patients around the time of laparoscopic surgery. Currently, I believe the laparoscopic TAP block is a valuable, yet underutilized tool in the field of Minimally Invasive Surgery.

i. Limitations:

1. Liposomal bupivacaine is a milky white color and it would have been very difficult to blind the surgeons infiltrating it as opposed to a placebo.
2. There is a learning curve with developing an ability to do the TAP block laparoscopically, however this technique has now been well practiced by our team.
3. BMI, additional procedures, history of other pain issues, such as fibromyalgia, may all be confounders to this study. All of these will be documented and hopefully averaged in the randomization.

VII. RISKS/BENEFITS

1. Risks and side effects related to the TAP Block with liposomal bupivacaine include bruising at the site of the injections, soreness, and a rare potential for intravascular injection causing cardiac arrhythmia. These risks are similar to the risk of routine bupivacaine in the trocar sites routinely used anyway. Of note, there were no complications of laparoscopic TAP blocks during the course of our recent trial #14-132.
2. There are no known direct benefits to study subjects.
3. If the study demonstrates a benefit of the TAP block in controlling post-operative pain better than simply using pre-incisional injections and decreases patient need for opiate analgesia this will undoubtedly benefit patients in future.
4. There are no potential ethical concerns with this study, especially given that it will be randomized.

BUDGET Primary costs incurred will be files and paper products for VAS scores, charting on recovery and post-op questionnaires. The cost of the procedural medications will be rolled into the global surgical charge as pre-incisional anesthetics are already routinely billed for.

RESEARCH ENVIRONMENT All procedures will all take place at the time of surgery in the operating room. Patients will receive information on the study in pre-op consultation or at the time of arrival to the Pre-op arena.

ELIGIBILITY:
Inclusion Criteria:

1. adult women
2. undergoing laparoscopic robotic assisted laparoscopic hysterectomy with or without removal of adnexa
3. Simultaneous procedures such as appendectomy, excision of endometriosis or pelvic lymph node dissection not an exclusion

Exclusion Criteria:

1. < 18
2. Not undergoing laparoscopic hysterectomy

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Gynecologic procedure applicable to females only.
Enrollment: 32 (Actual)
Dates: Start 2016-01-27 (Actual); Primary Completion 2017-04-15 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
Overall Benefit of Anesthesia Score (OBAS) | Post operative day 7
  Change in resting pain, vomiting, itching, sweating, freezing, dizziness, satisfaction Likert 0-10 0=not at all, 10- very much

SECONDARY OUTCOMES:
OBAS Questionnaire | Post operative day 1
  Changes in 7 measurements listed above
OBAS Questionnaire | Post operative day 2
  Changes in 7 measurements listed above

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] De Oliveira GS Jr, Milad MP, Fitzgerald P, Rahmani R, McCarthy RJ. Transversus abdominis plane infiltration and quality of recovery after laparoscopic hysterectomy: a randomized controlled trial. Obstet Gynecol. 2011 Dec;118(6):1230-1237. doi: 10.1097/AOG.0b013e318236f67f. PMID 22105251
- [Result] Jacobson GF, Shaber RE, Armstrong MA, Hung YY. Hysterectomy rates for benign indications. Obstet Gynecol. 2006 Jun;107(6):1278-83. doi: 10.1097/01.AOG.0000210640.86628.ff. PMID 16738152
- [Result] Committee opinion no. 628: robotic surgery in gynecology. Obstet Gynecol. 2015 Mar;125(3):760-767. doi: 10.1097/01.AOG.0000461761.47981.07. PMID 25730256
- [Result] Rafi AN. Abdominal field block: a new approach via the lumbar triangle. Anaesthesia. 2001 Oct;56(10):1024-6. doi: 10.1046/j.1365-2044.2001.02279-40.x. No abstract available. PMID 11576144
- [Result] Young MJ, Gorlin AW, Modest VE, Quraishi SA. Clinical implications of the transversus abdominis plane block in adults. Anesthesiol Res Pract. 2012;2012:731645. doi: 10.1155/2012/731645. Epub 2012 Jan 19. PMID 22312327
- [Result] Bhattacharjee S, Ray M, Ghose T, Maitra S, Layek A. Analgesic efficacy of transversus abdominis plane block in providing effective perioperative analgesia in patients undergoing total abdominal hysterectomy: A randomized controlled trial. J Anaesthesiol Clin Pharmacol. 2014 Jul;30(3):391-6. doi: 10.4103/0970-9185.137274. PMID 25190950
- [Result] Atim A, Bilgin F, Kilickaya O, Purtuloglu T, Alanbay I, Orhan ME, Kurt E. The efficacy of ultrasound-guided transversus abdominis plane block in patients undergoing hysterectomy. Anaesth Intensive Care. 2011 Jul;39(4):630-4. doi: 10.1177/0310057X1103900415. PMID 21823381